CLINICAL TRIAL: NCT00076141
Title: CSP #499A - Selenium and Vitamin E Cancer Prevention Trial - COHORT
Brief Title: Relatively Healthy Male Veterans Observed Over Time to See What Types of Diseases Develop
Acronym: ACTIVE Health
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 499A
Record Dates: First submitted 2004-01-14; First posted 2004-01-16 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: relatively healthy male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PE and buffy coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Older, Racially Diverse Males: Racially Divers Males over 50, expected to live more than 5 years

SUMMARY:
The purpose of this study is to gather a mixed racial group of relatively healthy male Veterans (for example, White, African-American, and Hispanic), who are at least 50 years of age. These men will be followed to see what types of diseases they develop and to determine if racial differences in lifestyle, blood test results, or genes are related to the types of diseases that are found. Diseases of particular interest are prostate cancer, other cancers, cardiovascular disease (for example, heart attacks and stroke), high blood pressure and diabetes. The group to be followed will consist of about 16,000 men recruited from about 40 VA Medical Centers across the country. Each man will be followed for at least five years depending on when he enters the study.

DETAILED DESCRIPTION:
The purpose of this study is to gather a mixed racial group of relatively healthy male Veterans (for example, White, African-American, and Hispanic), who are at least 50 years of age. These men will be followed to see what types of diseases they develop and to determine if racial differences in lifestyle, blood test results, or genes are related to the types of diseases that are found. Diseases of particular interest are prostate cancer, other cancers, cardiovascular disease (for example, heart attacks and stroke), high blood pressure and diabetes. The group to be followed will consist of about 16,000 men recruited from about 40 VA Medical Centers across the country. Each man will be followed for at least five years depending on when he enters the study.

Participants are asked to complete a set of forms to provide a brief medical history, demographics, information on lifestyle such as physical activities, smoking, and drinking, information on diet, and information on quality of life.

Subjects will be seen on a biannual basis with follow-up telephone interviews conducted during the intervening years. Follow-up telephone interviews will be conducted at the MAVERIC Call Center while follow-up clinic visits will take place at each SELECT site. In addition, VA clinical and administrative databases will be used to augment follow-up and confirm reported events.

During follow-up visits, participants will be asked whether they experienced any medical events since the last study visit, with information on specific diagnoses including prostate cancer, lung cancer, colon cancer, other cancers, stroke, myocardial infarction, hypertension, diabetes mellitus, kidney disease, chronic prostatitis, and benign prostatic hypertrophy. Confirmation of self-reported diagnosis will be made by an examination of discharge summaries, medical records, and available diagnostic and laboratory information by an end-points committee.

Recruitment for this observational cohort will proceed in parallel with recruitment for SELECT and can use SELECT staff and resources with very little additional burden in cost or staff time.

ELIGIBILITY:
Inclusion Criteria:

* relatively healthy male Veterans
* at least 50 years old

Exclusion Criteria:

* Life expectancy of at least 5 yrs

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — * relatively healthy male Veterans
  * at least 50 years old
Study Population: * relatively healthy male Veterans
  * at least 50 years old
Sampling Method: Non-Probability Sample
Enrollment: 991 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Chronic Conditions in African American and White Male Veterans | Every six months for at least five years
  To determine whether differences in the prevalence of common chronic conditions affecting older Veterans among African-American and white male Veterans are explained by medical, lifestyle, dietary, or other risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Gaziano, MD MPH, Study Chair — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (9):
- United States (9):
  - VA Medical Center, Loma Linda, Loma Linda, California
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Kansas City MO, Kansas City, Missouri
  - VA Medical Center, Northport, Northport, New York
  - VA Medical Center, Syracuse, Syracuse, New York
  - James H. Quillen VA Medical Center, Mountain Home, Tennessee
  - VA Medical Center, Huntington, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No